CLINICAL TRIAL: NCT06439823
Title: Controlled Study of Upper and Lower Limb Movements in Patients Patients with Pathologies That Have an Impact on Ambulation or Motor Function to Validate Signal Analysis Algorithms for Wearable Devices Using Magneto-inertial Technology
Brief Title: Controlled Study of Upper and Lower Limb Movements in Patients Patients with Pathologies That Have an Impact on Ambulation or Motor Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laurent Servais (Other)
Collaborators: SYSNAV (Industry)
Responsible Party: Sponsor-Investigator, Laurent Servais, Professor Laurent Servais, Centre Hospitalier Universitaire de Liege
Organization: Centre Hospitalier Universitaire de Liege (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MoCAP
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with neuromuscular disease or control subjects (Experimental): Patients and controls will be examined by a neuropediatric or neurologist. they will perform upper and lower limb assessments in a walking laboratory. this study comprises a single session per patient/control subject.
  Interventions: Device: ActiMyo®/Syde®

INTERVENTIONS:
Device: ActiMyo®/Syde® — Subjects will be equipped with magneto-inertial sensors (ActiMyo®/Syde®) and passive reflective markers belonging to the MoCap® motion capture system.

SUMMARY:
The main aim of the study is to validate the algorithms developed to analyze the signals from the various sensors contained in the magneto-inertial control units and reconstruct upper and lower limb movements under different normal and pathological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 2 years old
* Male or female
* Control subjects with no pathologies that have an impact on ambulation or motor function.
* Signed informed consent and, in the case of minors, informed consent signed by the person with parental authority/guardian

Exclusion Criteria:

* Any other previous or present pathology having an impact on current motor or balance function
* Recent surgery or trauma to upper or lower limbs, or major surgery or trauma within 6 months of inclusion.
* For control subjects, athlete of at least national level.
* Pregnant or breast-feeding women

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
step length and distance | 36 months
  Validate the algorithms developed to analyze the signals from the various sensors contained in magneto-inertial control units and reconstruct upper and lower limb movements.

CONTACTS AND LOCATIONS:
Locations (1):
- CHR citadelle, Liège, Liege, Belgium

IPD SHARING:
Plan to Share IPD: No